CLINICAL TRIAL: NCT03296696
Title: Phase 1/1b Study to Evaluate Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of AMG 596 as Monotherapy and in Combination With AMG 404 in Subjects With Glioblastoma or Malignant Glioma Expressing Mutant Epidermal Growth Factor Receptor Variant III (EGFRvIII)
Brief Title: Study of AMG 596 in Patients With EGFRvIII Positive Glioblastoma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Amgen business decision
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 20160132; 2017-001658-32 (EudraCT Number)
Record Dates: First submitted 2017-09-18; First posted 2017-09-28 (Actual); Results first posted 2024-10-29 (Actual); Last update posted 2024-10-29 (Actual); Status verified 2024-10

CONDITIONS: Glioblastoma or Malignant Glioma
Keywords: Phase 1/1b; EGFRvIII-positive glioblastoma or malignant glioma; safety and tolerability; AMG 596
MeSH Terms: conditions — Glioblastoma; Glioma

STUDY DESIGN:
Intervention Model Description: Bayesian logistic regression model
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Dose exploration (Experimental): Dose exploration of the intervention, AMG 596 alone or in combination with AMG 404
  Interventions: Drug: AMG 596; Drug: AMG 404
- Dose expansion (Experimental): Dose expansion of the intervention, AMG 596 alone or in combination with AMG 404
  Interventions: Drug: AMG 596; Drug: AMG 404

INTERVENTIONS:
Drug: AMG 596 — Drug
Drug: AMG 404 — Drug

SUMMARY:
This is a Phase 1/1b Study to Evaluate Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of AMG 596 monotherapy or in combination with AMG 404 in Subjects with Glioblastoma or Malignant Glioma Expressing Mutant Epidermal Growth Factor Receptor Variant III (EGFRvIII).

This is a first in human (FIH), open-label, sequential-dose-escalation study in subjects with EGFRvIII-positive glioblastoma or malignant glioma. This study will enroll 2 groups of subjects according to disease stage, recurrent disease (Group 1) and maintenance treatment after SoC in newly diagnosed disease (Group 2).

ELIGIBILITY:
Inclusion Criteria

* Eastern Cooperative Oncology Group (ECOG, Appendix G) Performance Status of less than or equal to 1
* Life expectancy of at least 3 months, in the opinion of the investigator.
* Must have pathologically documented, and definitively diagnosed World Health Organization (WHO) grade 4, glioblastoma or lower grade malignant gliomas with epidermal growth factor receptor variant III (EGFRvIII) positive tumor
* Must have recurrent disease confirmed by magnetic resonance imaging (MRI) (Group 1) or completed standard of care (SoC) therapy such as surgery with adjuvant radiochemotherapy with or without maintenance temozolomide according to local standards for newly diagnosed disease (Group 2)
* Hematological function as follows:

  * Absolute neutrophil count (ANC) greater than 1500/mm3 (1.5 × 10 9/L)
  * Platelet count greater than 100,000 mm3 (100 × 10 9/L)
  * White blood cell (WBC) count greater than 3 × 10 9/L
  * Hemoglobin greater than 9.0 g/dL
* Renal function as follows: serum creatinine less than 2.0 mg/dL and estimated glomerular filtration rate greater than or equal to 60 mL/min/1.73 m2 by Modification of Diet in Renal Disease (MDRD) and urine protein quantitative value of less than 30 mg/dL in urinalysis or less than or equal to 1+ on dipstick
* Hepatic function as follows:

  * Aspartate aminotransferase (AST) and Alanine aminotransferase (ALT) less than or equal to 3.0 x upper limit of normal (ULN)
  * Bilirubin less than or equal to 1.5 x ULN (unless considered due to Gilbert's syndrome or hemolysis)

Exclusion Criteria

* History or evidence of central nervous system bleeding as defined by stroke or intraocular bleed (including embolic stroke) not associated with any antitumor surgery within 6 months before enrolment
* Evidence of acute intracranial / intratumoral hemorrhage, except for subjects with stable grade 1 hemorrhage or fresh biopsy
* Known hypersensitivity to immunoglobulins or to any other component of the investigational product (IP) formulation
* Prior malignancy (other than in situ cancer) unless treated with curative intent and without evidence of disease for > 2 years before screening
* Active infection requiring intravenous antibiotics that was completed less than 1 week of study enrolment (day 1) with the exemption of prophylactic antibiotics for long line insertion or biopsy
* Known positive test for human immunodeficiency virus (HIV)
* Active hepatitis B and C based on the following results:

  * Positive for hepatitis B surface antigen (HepBsAg) (indicative of chronic hepatitis B or recent acute hepatitis B)
  * Negative HepBsAg and positive for hepatitis B core antibody: hepatitis B virus deoxyribonucleic acid (DNA) by polymerase chain reaction (PCR) is necessary. Detectable hepatitis B virus DNA suggests occult hepatitis B
  * Positive hepatitis C virus antibody (HepCAb): hepatitis C virus ribonucleic acid (RNA) by PCR is necessary. Detectable hepatitis C virus RNA suggests chronic hepatitis C Common terminology criteria for adverse events
* Unresolved toxicities from prior antitumor therapy, defined as not having resolved to common terminology criteria for adverse events (CTCAE), version 4.0 grade 1 (with the exception of myelosuppression, eg, neutropenia, anemia, thrombocytopenia), or to levels dictated in the eligibility criteria with the exception of alopecia or toxicities from prior antitumor therapy that are considered irreversible (defined as having been present and stable for greater than 2 months) which may be allowed if they are not otherwise described in the exclusion criteria AND there is agreement to allow by both the investigator and sponsor
* Antitumor therapy (chemotherapy, antibody therapy, molecular-targeted therapy, or investigational agent) within 14 days (Group 2 subjects) or 5 half-lives (whichever is longer: for Group 1 subjects) of day 1. Avastin, Pembrolizumab must be stopped 14 days prior to day 1
* Treatment with non-topical systemic corticosteroids within 14 days before enrollment (day 1) (exemption: prophylactic treatment with dexamethasone as defined in section 6.5, and systemic corticosteroid doses of ≤ 2 mg of dexamethasone (or equivalent) per day after consultation with Sponsor,)
* Prior participation in an investigational study (drug, procedure or device) within 21 days of study day 1
* Major surgery within 7 days of study day 1 with the exception of biopsy and long line insertion
* History or evidence of any other clinically significant disorder, condition or disease that, in the opinion of the investigator or Amgen physician, if consulted, would pose a risk to subject safety or interfere with the study evaluation, procedures or completion
* Male and female of reproductive potential who are unwilling to practice highly effective method(s) of birth control while on study and through 30 days after receiving the last dose of AMG 596 and through 4 months (120 days) after receiving the last dose of AMG 404.

  * Criteria for women of non-reproductive potential is as follows:
  * Postmenopausal as defined as:
  * Age of 55 years with cessation of menses for 12 months or more, OR
  * Age < 55 years and no spontaneous menses for at least 2 years, OR
  * Age < 55 years and spontaneous menses within the past year, but currently amenorrheic (eg, spontaneous or secondary to chemotherapy) AND with postmenopausal gonadotropin levels (luteinizing hormone and follicle-stimulating hormone level > 40 IU/L) or postmenopausal estradiol levels (< 5 ng/dL) according to the definition of "postmenopausal range" for the laboratory involved; OR
  * History of hysterectomy; OR
  * History of bilateral oophorectomy
  * Highly effective methods of birth control include sexual abstinence (male, female); vasectomy; bilateral tubal ligation/occlusion; hormonal birth control or intrauterine device (IUD) (female).
* Female who is lactating/breastfeeding or who plans to breastfeed while on study through 30 days after receiving the last dose of AMG 596 and through 4 months (120 days) after receiving the last dose of AMG 404.
* Female with a positive pregnancy test.
* Female planning to become pregnant while on study through 30 days after receiving the last dose of AMG 596 and through 4 months (120 days) after receiving the last dose of AMG 404 infusion.
* Male who is unwilling to abstain from sperm donation while on study through 30 days after receiving the last dose of AMG 596 and through 4 months (120 days) after receiving the last dose of AMG 404.
* Subjects likely to not be available to complete all protocol required study visits or procedures, and/or to comply with all required study procedures to the best of the subject and investigator's knowledge.
* History of solid organ transplantation. Prior treatment with anti-PD-1, anti-PD-L1, CTLA-4 or other checkpoint inhibitor drugs
* Prior treatment with AMG 596 monotherapy arm is not eligible to enroll in the combination therapy arm.
* Live vaccine therapies within 4 weeks prior to study drug administration
* Evidence of interstitial lung disease or active, non-infectious pneumonitis
* History of any immune-related colitis. Infectious colitis is allowed if evidence of adequate treatment and clinical recovery exists and at least 3 months interval observed since diagnosis of colitis.
* Active or history of any autoimmune disease or immunodeficiencies. Subjects with Type I diabetes, vitiligo, psoriasis, hypo-or hyper-thyroid disease not requiring immune-suppressive treatment are permitted.
* Myocardial infarction within 6 months of study day 1, symptomatic congestive heart failure (New York Heart Association > class II), unstable angina, or cardiac arrhythmia requiring medication.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-04-18 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2021-08-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (10):
- United States (2):
  - University of California Los Angeles, Los Angeles, California
  - Memorial Sloan Kettering Cancer Center, New York, New York
- Australia (2):
  - Royal North SHore Hospital, St Leonards, New South Wales
  - Peter MacCallum Cancer Centre, Melbourne, Victoria
- Gustave Roussy, Villejuif, France
- Germany (3):
  - UniversitÃ¤tsklinikum Carl Gustav Carus der Technischen UniversitÃ¤t Dresden, Dresden
  - Universitatsklinikum Hamburg-Eppendorf, Hamburg
  - Universitaetsklinikum Wuerzburg, WÃ¼rzburg
- Vrije Universiteit Medisch Centrum, Amsterdam, Netherlands
- Hospital Universitari Germans Trias i Pujol, Badalona, CataluÃ±a, Spain

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication (or other new use) have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors, and if not approved, may be further arbitrated by a Data Sharing Independent Review Panel. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the URL below.
URL: https://www.amgen.com/datasharing

REFERENCES:
- [Background] Sternjak A, Lee F, Thomas O, Balazs M, Wahl J, Lorenczewski G, Ullrich I, Muenz M, Rattel B, Bailis JM, Friedrich M. Preclinical Assessment of AMG 596, a Bispecific T-cell Engager (BiTE) Immunotherapy Targeting the Tumor-specific Antigen EGFRvIII. Mol Cancer Ther. 2021 May;20(5):925-933. doi: 10.1158/1535-7163.MCT-20-0508. Epub 2021 Feb 25. PMID 33632870
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled from April 18, 2018 and last participant visit was August 28, 2021. Participants enrolled at 9 centers in United States, Australia, France, Germany, Netherlands, and Spain.
Pre-assignment Details: Of the planned 200 participants, 30 were enrolled. Of the 30 participants enrolled, 29 received investigational product. Due to early termination, participants were only enrolled into dose escalation AMG 596 monotherapy arms.
Groups:
- AMG 596 Monotherapy 4.5 mcg: Participants received 4.5 mcg of AMG 596 by continuous intravenous (cIV) infusion on a 7-days on/7-days off dosing schedule until treatment discontinuation criteria were applied.
- AMG 596 Monotherapy 15 mcg: The first participant received 15 mcg of AMG 596 by cIV infusion on a 7-days on/7-days off dosing schedule until treatment discontinuation criteria were applied. The remaining 2 participants received 15 mcg of AMG 596 by cIV infusion on a 28-days on/14-days off dosing schedule until treatment discontinuation criteria were applied.
- AMG 596 Monotherapy 45 mcg: Participants received 45 mcg of AMG 596 by cIV infusion on a 28-days on/14-days off dosing schedule until treatment discontinuation criteria were applied.
- AMG 596 Monotherapy 150 mcg: Participants received 150 mcg of AMG 596 by cIV infusion on a 28-days on/14-days off dosing schedule until treatment discontinuation criteria were applied.
- AMG596 Monotherapy 500 mcg: Participants received 500 mcg of AMG 596 by cIV infusion on a 28-days on/14-days off dosing schedule until treatment discontinuation criteria were applied.
- AMG596 Monotherapy 1000 mcg: Participants received 1000 mcg of AMG 596 by cIV infusion on a 28-days on/14-days off dosing schedule until treatment discontinuation criteria were applied.
- AMG596 Monotherapy 1500 mcg: Participants received 1500 mcg of AMG 596 by cIV infusion on a 28-days on/14-days off dosing schedule until treatment discontinuation criteria were applied.
- AMG596 Monotherapy 3000 mcg: Participants received 3000 mcg of AMG 596 by cIV infusion on a 28-days on/14-days off dosing schedule until treatment discontinuation criteria were applied.
- AMG596 Monotherapy 6000 mcg: Participants received 6000 mcg of AMG 596 by cIV infusion on a 7-days on/7-days off dosing schedule until treatment discontinuation criteria were applied.
- AMG596 Monotherapy 1500/15 mcg: The participant was enrolled into AMG 596 Monotherapy 15 mcg cIV infusion arm but received an overdose (1500 mcg). Based on Food and Drug Administration recommendation, the participant received 1500 mcg/day during Week 1, followed by 15 mcg/day during Weeks 2 to 4, followed by a 2-week break.
Period: Overall Study
Arm/Group | AMG 596 Monotherapy 4.5 mcg | AMG 596 Monotherapy 15 mcg | AMG 596 Monotherapy 45 mcg | AMG 596 Monotherapy 150 mcg | AMG596 Monotherapy 500 mcg | AMG596 Monotherapy 1000 mcg | AMG596 Monotherapy 1500 mcg | AMG596 Monotherapy 3000 mcg | AMG596 Monotherapy 6000 mcg | AMG596 Monotherapy 1500/15 mcg
Started | 1 | 3 | 3 | 4 | 4 | 4 | 4 | 5 | 1 | 1
Received Investigational Product | 1 | 3 | 3 | 4 | 3 | 4 | 4 | 5 | 1 | 1
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not Completed | 1 | 3 | 3 | 4 | 4 | 4 | 3 | 5 | 1 | 1
Not completed — Started Other Antitumor Therapy | 1 | 2 | 1 | 2 | 1 | 1 | 2 | 3 | 1 | 0
Not completed — Death | 0 | 1 | 1 | 2 | 2 | 3 | 1 | 2 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Baseline data were collected for all enrolled participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | AMG 596 Monotherapy 4.5 mcg | AMG 596 Monotherapy 15 mcg | AMG 596 Monotherapy 45 mcg | AMG 596 Monotherapy 150 mcg | AMG596 Monotherapy 500 mcg | AMG596 Monotherapy 1000 mcg | AMG596 Monotherapy 1500 mcg | AMG596 Monotherapy 3000 mcg | AMG596 Monotherapy 6000 mcg | AMG596 Monotherapy 1500/15 mcg | Total
Number analyzed (Participants) | 1 | 3 | 3 | 4 | 4 | 4 | 4 | 5 | 1 | 1 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 1 | 3 | 3 | 3 | 3 | 4 | 4 | 5 | 1 | 1 | 28
  >=65 years | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 2
Age, Continuous [Mean (Standard Deviation); unit: Years] | 62.0 (NA) — Standard deviation cannot be calculated for a single participant. | 51.0 (6.1) | 56.7 (8.7) | 58.0 (7.5) | 51.5 (13.6) | 55.0 (4.9) | 51.5 (12.4) | 53.0 (5.5) | 44.0 (NA) — Standard deviation cannot be calculated for a single participant. | 49.0 (NA) — Standard deviation cannot be calculated for a single participant. | 54.1 (7.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 0 | 2 | 1 | 1 | 1 | 0 | 1 | 1 | 10
  Male | 0 | 1 | 3 | 2 | 3 | 3 | 3 | 5 | 0 | 0 | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 1 | 3 | 3 | 4 | 3 | 4 | 4 | 5 | 1 | 1 | 29
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White | 1 | 2 | 3 | 4 | 3 | 3 | 4 | 2 | 1 | 1 | 24
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 3 | 0 | 0 | 4

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose-Limiting Toxicities (DLTs)
Description: A DLT was any of the following occurring and regarded by the investigator as related to AMG 596. Hematological DLTs: absolute neutrophil count (ANC) <0.5×10^9/L for ≥7 days, febrile neutropenia with ANC<0.5×10^9/L and fever ≥38.5°C, platelets<50×10^9/L>7 days or clinically significant bleeding. Non-hematological DLTs: any grade 4 non-hematological toxicity, any grade ≥3 non-hematological toxicity if nausea and vomiting, grade 3 non-hematologic toxicity lasting >3 days despite treatment, grade 3 fatigue wasn't classified as DLT, grade 3 acute kidney injury, grade 3 seizure, ataxia, encephalopathy, other grade 3 neurologic-related adverse events lasting >3 days despite treatment, neurologic-related adverse event leading to treatment interruption needing>1 week to resolve to grade≤1, any grade 3 endocrinopathy that can't be controlled by hormonal replacement. Toxicity grading was graded using the Common Terminology Criteria for Adverse Events (CTCAE v4.0)
Time Frame: Up to 28 days
Population: The DLT Evaluable Analysis Set included all participants in the 7-day on/7-day off dosing groups who completed 100% of planned doses and all participants in the 28-day on/14-day off dosing groups who completed 90% of planned doses.
Measure: Count of Participants; unit: Participants
Arm/Group | AMG 596 Monotherapy 4.5 mcg | AMG 596 Monotherapy 15 mcg | AMG 596 Monotherapy 45 mcg | AMG 596 Monotherapy 150 mcg | AMG596 Monotherapy 500 mcg | AMG596 Monotherapy 1000 mcg | AMG596 Monotherapy 1500 mcg | AMG596 Monotherapy 3000 mcg | AMG596 Monotherapy 6000 mcg | AMG596 Monotherapy 1500/15 mcg
Number analyzed (Participants) | 1 | 3 | 3 | 4 | 3 | 4 | 4 | 5 | 1 | 1
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

2. Primary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs)
Description: An adverse event (AE) was defined as any untoward medical occurrence in a clinical trial participant. A TEAE was any AE that begun or worsened after the initial dose of investigational product. Any clinically significant changes in vital signs, physical examinations, and clinical laboratory tests that begun or worsened after the initial dose of investigational product were recorded as TEAEs.
Time Frame: First dose of study drug until 37 days after last dose or end of study, whichever is earlier. Duration with median (min, max) in months: 3.32 (1.28, 29.31)
Population: The safety analysis set included all participants who were enrolled and received at least 1 dose of AMG 596.
Measure: Count of Participants; unit: Participants
Arm/Group | AMG 596 Monotherapy 4.5 mcg | AMG 596 Monotherapy 15 mcg | AMG 596 Monotherapy 45 mcg | AMG 596 Monotherapy 150 mcg | AMG596 Monotherapy 500 mcg | AMG596 Monotherapy 1000 mcg | AMG596 Monotherapy 1500 mcg | AMG596 Monotherapy 3000 mcg | AMG596 Monotherapy 6000 mcg | AMG596 Monotherapy 1500/15 mcg
Number analyzed (Participants) | 1 | 3 | 3 | 4 | 3 | 4 | 4 | 5 | 1 | 1
Participants | 1 | 3 | 3 | 4 | 3 | 3 | 4 | 5 | 1 | 1

3. Primary Outcome: Number of Participants With Treatment-Related Adverse Events (AEs)
Description: A treatment-related AE was defined as any untoward medical occurrence in a clinical trial participant that was considered related to the investigational product. Any clinically significant changes in vital signs, physical examinations, and clinical laboratory tests that were considered related to the investigational product were recorded as treatment-related AEs.
Time Frame: as for outcome 2
Population: The safety analysis set included all participants who were enrolled and received at least 1 dose of AMG 596.
Measure: Count of Participants; unit: Participants
Arm/Group | AMG 596 Monotherapy 4.5 mcg | AMG 596 Monotherapy 15 mcg | AMG 596 Monotherapy 45 mcg | AMG 596 Monotherapy 150 mcg | AMG596 Monotherapy 500 mcg | AMG596 Monotherapy 1000 mcg | AMG596 Monotherapy 1500 mcg | AMG596 Monotherapy 3000 mcg | AMG596 Monotherapy 6000 mcg | AMG596 Monotherapy 1500/15 mcg
Number analyzed (Participants) | 1 | 3 | 3 | 4 | 3 | 4 | 4 | 5 | 1 | 1
Participants | 1 | 3 | 3 | 3 | 3 | 2 | 4 | 4 | 1 | 1

4. Secondary Outcome: Average Steady-state Concentration (Css) of Serum AMG 596
Time Frame: Cycle1 to Cycle2 (cycle=14 days in single participant cohorts,42 days in multiple participant cohorts):7-days on/7-days off dosing and 28-days on/14-days off dosing:pre-infusion,2,6,8,24,48hrs post-infusion start,0.5,2,4,8,24hrs post infusion end
Population: The pharmacokinetic (PK) analysis set contained all participants who received the investigational product and had available PK data for each timepoint.
Measure: Mean (Full Range); unit: ng/mL
Arm/Group | AMG 596 Monotherapy 4.5 mcg | AMG 596 Monotherapy 15 mcg | AMG 596 Monotherapy 45 mcg | AMG 596 Monotherapy 150 mcg | AMG596 Monotherapy 500 mcg | AMG596 Monotherapy 1000 mcg | AMG596 Monotherapy 1500 mcg | AMG596 Monotherapy 3000 mcg | AMG596 Monotherapy 6000 mcg | AMG596 Monotherapy 1500/15 mcg
Number analyzed (Participants) | 1 | 3 | 3 | 4 | 3 | 4 | 4 | 5 | 1 | 1
ng/mL
  Cycle 1: number analyzed (Participants) | 1 | 2 | 3 | 4 | 3 | 4 | 4 | 5 | 1 | 1
  Cycle 1 | 0.733 [0.733 to 0.733] | 1.90 [1.87 to 1.93] | 3.38 [3.28 to 3.47] | 9.53 [2.98 to 14.0] | 26.7 [22.4 to 29.8] | 67.1 [45.9 to 89.0] | 106 [72.5 to 136] | 180 [103 to 222] | 610 [610 to 610] | 19.4 [19.4 to 19.4]
  Cycle 2: number analyzed (Participants) | 1 | 3 | 2 | 3 | 2 | 3 | 3 | 3 | 1 | 0
  Cycle 2 | 0.548 [0.548 to 0.548] | 1.48 [0.872 to 2.51] | 3.37 [2.81 to 3.93] | 11.4 [6.91 to 13.7] | 36.2 [25.6 to 46.9] | 74.3 [25.0 to 144] | 115 [60.1 to 157] | 194 [148 to 254] | 807 [807 to 807] |

5. Secondary Outcome: Area Under the Concentration-time Curve (AUC) for Serum AMG 596
Description: There were insufficient evaluable samples collected for the determination of AUC.
Time Frame: as for outcome 4
Population: The pharmacokinetic (PK) analysis set contained all participants who received the investigational product and had available PK data for each timepoint. 0 participants had evaluable data for the determination of AUC, therefore 0 participants were analyzed for this endpoint.
Arm/Group | AMG 596 Monotherapy 4.5 mcg | AMG 596 Monotherapy 15 mcg | AMG 596 Monotherapy 45 mcg | AMG 596 Monotherapy 150 mcg | AMG596 Monotherapy 500 mcg | AMG596 Monotherapy 1000 mcg | AMG596 Monotherapy 1500 mcg | AMG596 Monotherapy 3000 mcg | AMG596 Monotherapy 6000 mcg | AMG596 Monotherapy 1500/15 mcg
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

6. Secondary Outcome: Clearance for Serum AMG 596
Description: Clearance (CL) is calculated based on dose and AUC.
Time Frame: as for outcome 4
Population: as for outcome 4
Measure: Mean (Full Range); unit: mcg/day/(hr*ng/mL)
Arm/Group | AMG 596 Monotherapy 4.5 mcg | AMG 596 Monotherapy 15 mcg | AMG 596 Monotherapy 45 mcg | AMG 596 Monotherapy 150 mcg | AMG596 Monotherapy 500 mcg | AMG596 Monotherapy 1000 mcg | AMG596 Monotherapy 1500 mcg | AMG596 Monotherapy 3000 mcg | AMG596 Monotherapy 6000 mcg | AMG596 Monotherapy 1500/15 mcg
Number analyzed (Participants) | 1 | 2 | 3 | 3 | 3 | 4 | 4 | 4 | 1 | 1
mcg/day/(hr*ng/mL)
  Cycle 1 | 0.0324 [0.0324 to 0.0324] | 0.0116 [0.0102 to 0.0130] | 0.0172 [0.0122 to 0.0200] | 0.0207 [0.0161 to 0.0294] | 0.0272 [0.0244 to 0.0309] | 0.0237 [0.0188 to 0.0322] | 0.0218 [0.0171 to 0.0308] | 0.0291 [0.0197 to 0.0464] | 0.0146 [0.0146 to 0.0146] | 0.158 [0.158 to 0.158]
  Cycle 2: number analyzed (Participants) | 1 | 2 | 1 | 3 | 0 | 1 | 2 | 1 | 1 | 0
  Cycle 2 | 0.0469 [0.0469 to 0.0469] | 0.0175 [0.00910 to 0.0259] | 0.0232 [0.0232 to 0.0232] | 0.0228 [0.0163 to 0.0309] |  | 0.0256 [0.0256 to 0.0256] | 0.0161 [0.0147 to 0.0175] | 0.0245 [0.0245 to 0.0245] | 0.0113 [0.0113 to 0.0113] |

7. Secondary Outcome: Apparent Volume of Distribution at Steady-State for Serum AMG 596
Description: The formula for volume of distribution is dose/concentration. For this study, the dose is measured in mcg/day and concentration is measure as ng/mL resulting in units of mcg/day/(ng/mL) for volume of distribution.
Time Frame: as for outcome 4
Population: as for outcome 4
Measure: Mean (Full Range); unit: mcg/day/(ng/mL)
Arm/Group | AMG 596 Monotherapy 4.5 mcg | AMG 596 Monotherapy 15 mcg | AMG 596 Monotherapy 45 mcg | AMG 596 Monotherapy 150 mcg | AMG596 Monotherapy 500 mcg | AMG596 Monotherapy 1000 mcg | AMG596 Monotherapy 1500 mcg | AMG596 Monotherapy 3000 mcg | AMG596 Monotherapy 6000 mcg | AMG596 Monotherapy 1500/15 mcg
Number analyzed (Participants) | 1 | 2 | 3 | 3 | 3 | 4 | 4 | 4 | 1 | 1
mcg/day/(ng/mL)
  Cycle 1 | 0.269 [0.269 to 0.269] | 0.0961 [0.0637 to 0.128] | 0.173 [0.125 to 0.213] | 0.247 [0.198 to 0.325] | 0.200 [0.155 to 0.280] | 0.212 [0.109 to 0.278] | 0.205 [0.155 to 0.268] | 0.269 [0.185 to 0.387] | 0.166 [0.166 to 0.166] | 1.61 [1.61 to 1.61]
  Cycle 2: number analyzed (Participants) | 1 | 2 | 1 | 3 | 0 | 1 | 2 | 1 | 1 | 0
  Cycle 2 | 0.289 [0.289 to 0.289] | 0.162 [0.0929 to 0.232] | 0.246 [0.246 to 0.246] | 0.242 [0.158 to 0.354] |  | 0.223 [0.223 to 0.223] | 0.140 [0.0836 to 0.196] | 0.235 [0.235 to 0.235] | 0.115 [0.115 to 0.115] |

8. Secondary Outcome: Terminal Half-life (t1/2) Associated With Lambda z (λz) for Serum AMG 596
Time Frame: as for outcome 4
Population: as for outcome 4
Measure: Mean (Full Range); unit: Hours
Arm/Group | AMG 596 Monotherapy 4.5 mcg | AMG 596 Monotherapy 15 mcg | AMG 596 Monotherapy 45 mcg | AMG 596 Monotherapy 150 mcg | AMG596 Monotherapy 500 mcg | AMG596 Monotherapy 1000 mcg | AMG596 Monotherapy 1500 mcg | AMG596 Monotherapy 3000 mcg | AMG596 Monotherapy 6000 mcg | AMG596 Monotherapy 1500/15 mcg
Number analyzed (Participants) | 1 | 2 | 3 | 3 | 3 | 4 | 4 | 4 | 1 | 1
Hours
  Cycle 1 | 5.75 [5.75 to 5.75] | 5.59 [4.34 to 6.84] | 6.98 [6.42 to 7.39] | 8.44 [7.66 to 9.10] | 5.02 [4.37 to 6.29] | 6.16 [3.96 to 7.49] | 6.67 [5.31 to 8.51] | 6.54 [5.77 to 7.23] | 7.90 [7.90 to 7.90] | 7.04 [7.04 to 7.04]
  Cycle 2: number analyzed (Participants) | 1 | 2 | 1 | 3 | 0 | 1 | 2 | 1 | 1 | 0
  Cycle 2 | 4.27 [4.27 to 4.27] | 6.64 [6.21 to 7.07] | 7.33 [7.33 to 7.33] | 7.23 [6.72 to 7.94] |  | 6.05 [6.05 to 6.05] | 5.87 [3.95 to 7.79] | 6.64 [6.64 to 6.64] | 7.05 [7.05 to 7.05] |

9. Secondary Outcome: Number of Participants With an Objective Response (OR) Per Modified Response Assessment in Neuro-Oncology Criteria (RANO) Criteria With AMG 596 Monotherapy
Description: Objective response was defined as the number of participants with complete response (CR) or partial response (PR) per modified RANO criteria. CR per modified RANO: disappearance of all enhancing disease, no new lesions, stable or improved T2-weighted fluid-attenuated inversion recovery (T2/FLAIR), no more than physiological steroids, clinically stable or improved, disappearance confirmed with follow-up scans after ≥4 weeks. PR per modified RANO: ≥50% decrease in the sum of perpendicular diameters of enhancing disease from baseline, stable or improved T2/FLAIR, stable or decreased steroid dose, clinically stable or improved, decrease confirmed with follow up scan after ≥ 4 weeks.
Time Frame: Baseline up to 12 Months
Population: The RANO Evaluable Analysis set included all participants that were enrolled and received at least one administration of AMG 596 and who had at least one measurable lesion identified by the Principal Investigator at baseline.
Measure: Count of Participants; unit: Participants
Arm/Group | AMG 596 Monotherapy 4.5 mcg | AMG 596 Monotherapy 15 mcg | AMG 596 Monotherapy 45 mcg | AMG 596 Monotherapy 150 mcg | AMG596 Monotherapy 500 mcg | AMG596 Monotherapy 1000 mcg | AMG596 Monotherapy 1500 mcg | AMG596 Monotherapy 3000 mcg | AMG596 Monotherapy 6000 mcg | AMG596 Monotherapy 1500/15 mcg
Number analyzed (Participants) | 1 | 3 | 3 | 4 | 3 | 4 | 3 | 5 | 1 | 1
Participants | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

10. Secondary Outcome: Time to Response With AMG 596 Monotherapy
Description: Time to response was calculated as the number of months from the date of first administration of AMG 596 to the date of confirmation of first objective response per magnetic resonance imaging (MRI) scan. If a participant did not respond, time to response was censored at the date of the last evaluable response assessment.
Time Frame: Up to 12 months
Population: The safety analysis set included all participants who were enrolled and received at least 1 dose of AMG 596. Only participants with OR were used for this analysis.
Measure: Median (80% Confidence Interval); unit: Months
Arm/Group | AMG 596 Monotherapy 4.5 mcg | AMG 596 Monotherapy 15 mcg | AMG 596 Monotherapy 45 mcg | AMG 596 Monotherapy 150 mcg | AMG596 Monotherapy 500 mcg | AMG596 Monotherapy 1000 mcg | AMG596 Monotherapy 1500 mcg | AMG596 Monotherapy 3000 mcg | AMG596 Monotherapy 6000 mcg | AMG596 Monotherapy 1500/15 mcg
Number analyzed (Participants) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Months |  | 7.0 [NA to NA] — Only 1 participant with evaluable data, therefore lower and upper confidence intervals could not be calculated. |  |  |  |  |  |  |  |

11. Secondary Outcome: Response Duration With AMG 596 Monotherapy
Description: Response duration was analysed as the number of months between the first tumor response assessment of an OR (PR or CR) which is subsequently confirmed to the time of the first tumor response assessment of progressive disease or death if due to disease progression.
Time Frame: Up to 30 months
Population: as for outcome 10
Measure: Median (80% Confidence Interval); unit: Months
Arm/Group | AMG 596 Monotherapy 4.5 mcg | AMG 596 Monotherapy 15 mcg | AMG 596 Monotherapy 45 mcg | AMG 596 Monotherapy 150 mcg | AMG596 Monotherapy 500 mcg | AMG596 Monotherapy 1000 mcg | AMG596 Monotherapy 1500 mcg | AMG596 Monotherapy 3000 mcg | AMG596 Monotherapy 6000 mcg | AMG596 Monotherapy 1500/15 mcg
Number analyzed (Participants) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Months |  | 27.9 [NA to NA] — Only 1 participant with evaluable data, therefore lower and upper confidence intervals could not be calculated. |  |  |  |  |  |  |  |

12. Secondary Outcome: Time to Progression (TTP) With AMG 596 Monotherapy
Description: The TTP was calculated as the time from the date of first dose of AMG 596 until the date of diagnosis of progression of tumor. Participants who did not have progression were censored at the last radiological non-missing evaluable tumor assessment date.
Time Frame: Up to 12 Months
Population: The safety analysis set included all participants who were enrolled and received at least 1 dose of AMG 596
Measure: Median (80% Confidence Interval); unit: Months
Arm/Group | AMG 596 Monotherapy 4.5 mcg | AMG 596 Monotherapy 15 mcg | AMG 596 Monotherapy 45 mcg | AMG 596 Monotherapy 150 mcg | AMG596 Monotherapy 500 mcg | AMG596 Monotherapy 1000 mcg | AMG596 Monotherapy 1500 mcg | AMG596 Monotherapy 3000 mcg | AMG596 Monotherapy 6000 mcg | AMG596 Monotherapy 1500/15 mcg
Number analyzed (Participants) | 1 | 3 | 3 | 4 | 3 | 4 | 4 | 5 | 1 | 1
Months | 2.1 [NA to NA] — Only 1 participant in the treatment arm, therefore confidence intervals cannot be calculated. | 1.9 [0.7 to NA] — Values are not evaluable as the upper limit was not reached. | 1.9 [1.2 to NA] — Values are not evaluable as the upper limit was not reached. | 2.6 [2.4 to NA] — Values are not evaluable as the upper limit was not reached. | 1.2 [0.1 to NA] — Values are not evaluable as the upper limit was not reached. | 1.7 [1.0 to NA] — Values are not evaluable as the upper limit was not reached. | 2.4 [1.2 to NA] — Values are not evaluable as the upper limit was not reached. | 7.0 [1.3 to NA] — Values are not evaluable as the upper limit was not reached. | 5.3 [NA to NA] — Only 1 participant in the treatment arm, therefore confidence intervals cannot be calculated. | 2.6 [NA to NA] — Only 1 participant in the treatment arm, therefore confidence intervals cannot be calculated.

13. Secondary Outcome: Progression-free Survival (PFS) With AMG 596 Monotherapy
Description: The PFS was calculated as the time from the date of first dose of AMG 596 until the date of diagnosis of progression of tumor, or date of death, whichever was earlier.
Time Frame: Up to 12 months
Population: The safety analysis set included all participants who were enrolled and received at least 1 dose of AMG 596.
Measure: Median (80% Confidence Interval); unit: Months
Arm/Group | AMG 596 Monotherapy 4.5 mcg | AMG 596 Monotherapy 15 mcg | AMG 596 Monotherapy 45 mcg | AMG 596 Monotherapy 150 mcg | AMG596 Monotherapy 500 mcg | AMG596 Monotherapy 1000 mcg | AMG596 Monotherapy 1500 mcg | AMG596 Monotherapy 3000 mcg | AMG596 Monotherapy 6000 mcg | AMG596 Monotherapy 1500/15 mcg
Number analyzed (Participants) | 1 | 3 | 3 | 4 | 3 | 4 | 4 | 5 | 1 | 1
Months | 2.1 [NA to NA] — Only 1 participant in the treatment arm, therefore confidence intervals cannot be calculated. | 1.9 [0.7 to NA] — Upper confidence limit could not be calculated due to the low number of events reported. | 1.9 [1.2 to NA] — Upper confidence limit could not be calculated due to the low number of events reported. | 2.6 [2.4 to NA] — Upper confidence limit could not be calculated due to the low number of events reported. | 1.2 [0.1 to NA] — Upper confidence limit could not be calculated due to the low number of events reported. | 1.7 [1.0 to NA] — Upper confidence limit could not be calculated due to the low number of events reported. | 2.4 [1.2 to NA] — Upper confidence limit could not be calculated due to the low number of events reported. | 5.8 [1.3 to NA] — Upper confidence limit could not be calculated due to the low number of events reported. | 5.3 [NA to NA] — Only 1 participant in the treatment arm, therefore confidence intervals cannot be calculated. | 2.6 [NA to NA] — Only 1 participant in the treatment arm, therefore confidence intervals cannot be calculated.

ADVERSE EVENTS:
Time Frame: Mortality duration with median (min, max) in months: 4.27 (0.20, 35.48). Adverse Event duration with median (min, max) in months: 3.32 (1.28, 29.31).
Description: Serious and Other Adverse Events were collected for all participants who received at least one dose of study drug. All Cause Mortality was collected for all enrolled participants.
Groups:
- AMG596 4.5 mcg: AMG596 4.5 mcg/day 7 Day cIV
- AMG596 15 mcg: AMG596 15 mcg/day 7/28 Day cIV
- AMG596 45 mcg: AMG596 45 mcg/day 28 Day cIV
- AMG596 150 mcg: AMG596 150 mcg/day 28 Day cIV
- AMG596 500 mcg: AMG596 500 mcg/day 28 Day cIV
- AMG596 1000 mcg: AMG596 1000 mcg/day 28 Day cIV
- AMG596 1500 mcg: AMG596 1500 mcg/day 28 Day cIV
- AMG596 3000 mcg: AMG596 3000 mcg/day 28 Day cIV
- AMG596 6000 mcg: AMG596 6000 mcg/day 28 Day cIV
- AMG596 1500/15 mcg: AMG596 1500/15 mcg/day 28 Day cIV
Arm/Group | AMG596 4.5 mcg | AMG596 15 mcg | AMG596 45 mcg | AMG596 150 mcg | AMG596 500 mcg | AMG596 1000 mcg | AMG596 1500 mcg | AMG596 3000 mcg | AMG596 6000 mcg | AMG596 1500/15 mcg
All-Cause Mortality (participants affected / at risk) | 0/1 | 1/3 | 1/3 | 2/4 | 2/4 | 3/4 | 1/4 | 2/5 | 0/1 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1 | 3/3 | 1/3 | 3/4 | 2/3 | 2/4 | 3/4 | 3/5 | 1/1 | 1/1
Other Adverse Events (participants affected / at risk) | 1/1 | 3/3 | 3/3 | 4/4 | 3/3 | 3/4 | 4/4 | 5/5 | 1/1 | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | AMG596 4.5 mcg (N=1) | AMG596 15 mcg (N=3) | AMG596 45 mcg (N=3) | AMG596 150 mcg (N=4) | AMG596 500 mcg (N=3) | AMG596 1000 mcg (N=4) | AMG596 1500 mcg (N=4) | AMG596 3000 mcg (N=5) | AMG596 6000 mcg (N=1) | AMG596 1500/15 mcg (N=1)
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
General physical health deterioration (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hyperthermia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Catheter site infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Device related infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vascular access site infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Vascular device infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Wound infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Shunt malfunction (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Vascular access complication (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Glioblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Glioblastoma multiforme (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Aphasia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Depressed level of consciousness (Nervous system disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 1
Hydrocephalus (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Seizure (Nervous system disorders) | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 1 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | AMG596 4.5 mcg (N=1) | AMG596 15 mcg (N=3) | AMG596 45 mcg (N=3) | AMG596 150 mcg (N=4) | AMG596 500 mcg (N=3) | AMG596 1000 mcg (N=4) | AMG596 1500 mcg (N=4) | AMG596 3000 mcg (N=5) | AMG596 6000 mcg (N=1) | AMG596 1500/15 mcg (N=1)
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 1 | 0 | 1 | 1 | 0 | 1 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Lymphopenia (Blood and lymphatic system disorders) | 1 | 1 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Normocytic anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cushingoid (Endocrine disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Chalazion (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Eye disorder (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Lacrimation increased (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Visual acuity reduced (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Visual impairment (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Anal incontinence (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 1 | 1 | 1 | 0 | 0 | 0 | 2 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypoaesthesia oral (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 2 | 1 | 1 | 1 | 2 | 1 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1 | 2 | 1 | 0 | 1 | 0 | 0 | 1
Asthenia (General disorders) | 1 | 0 | 0 | 2 | 1 | 0 | 0 | 1 | 0 | 0
Catheter site thrombosis (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chest pain (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Chills (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Device related thrombosis (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 3 | 2 | 0 | 1 | 1 | 1 | 3 | 1 | 1
Gait disturbance (General disorders) | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0
Malaise (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Mucosal inflammation (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oedema (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 2 | 1 | 1 | 1 | 0 | 0 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cytokine release syndrome (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Immune system disorder (Immune system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Catheter site infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Device related infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Skin infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Urinary tract infection bacterial (Infections and infestations) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Urinary tract infection staphylococcal (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vascular device infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Viral infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Wound infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Vascular access complication (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Wound haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Alanine aminotransferase abnormal (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 0 | 0
Aspartate aminotransferase abnormal (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Blood bilirubin increased (Investigations) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
C-reactive protein increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 1
CD4 lymphocytes decreased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Interleukin level increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lipase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Lymphocyte count abnormal (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Lymphocyte count decreased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
White blood cell count decreased (Investigations) | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
White blood cell count increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Dyslipidaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperchloraemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0
Hypouricaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Metabolic disorder (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Amnesia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Aphasia (Nervous system disorders) | 0 | 1 | 0 | 2 | 2 | 2 | 0 | 1 | 0 | 0
Ataxia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0
Balance disorder (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Brain oedema (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cognitive disorder (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Depressed level of consciousness (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 1 | 0 | 1 | 1 | 1 | 1 | 0 | 0
Dysarthria (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dyskinesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dysmetria (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Epilepsy (Nervous system disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 1 | 2 | 2 | 2 | 2 | 2 | 3 | 4 | 0 | 1
Hemianopia homonymous (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hemiparesis (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 0 | 0
Hydrocephalus (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypersomnia (Nervous system disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypokinesia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Language disorder (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Lethargy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Memory impairment (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Neuropathy peripheral (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pyramidal tract syndrome (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Seizure (Nervous system disorders) | 0 | 1 | 1 | 1 | 1 | 0 | 0 | 2 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Device malfunction (Product Issues) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Bradyphrenia (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Confusional state (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Depressed mood (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Depression (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Disorientation (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bladder spasm (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Polyuria (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Urinary incontinence (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Blister (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Onychoclasis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Purpura (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 2 | 1 | 0 | 0 | 0
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Skin irritation (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Haematoma (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hot flush (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Hypotension (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Phlebitis superficial (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Thrombophlebitis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Thrombosis (Vascular disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0

LIMITATIONS AND CAVEATS:
The study was terminated early. Therefore, a smaller number of participants than planned were enrolled and analysed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.

DOCUMENTS (2):
  • Study Protocol (2019-07-29): https://cdn.clinicaltrials.gov/large-docs/96/NCT03296696/Prot_000.pdf
  • Statistical Analysis Plan (2019-05-20): https://cdn.clinicaltrials.gov/large-docs/96/NCT03296696/SAP_001.pdf